CLINICAL TRIAL: NCT03331237
Title: Shoulder Analgesia Sparing Diaphragm; ISO Block Versus Low Volume Scalene Block. A Randomized Controlled Double Blind Study
Brief Title: Sparing Diaphragm; ISO Block Versus Low Volume Scalene Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Healthpoint Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Muhammad Taha, Consultant of aneathesia, Healthpoint Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REC007
Record Dates: First submitted 2017-10-28; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Shoulder Arthropathy Associated With Other Conditions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LVS group (Active Comparator): interscalene injection
  Interventions: Procedure: scalene block
- ISO group (Active Comparator): in this group all patients will receive ISO block.
  Interventions: Procedure: ISO block

INTERVENTIONS:
Procedure: scalene block — scalene block using 5ml of ropivacaine
  Arms: LVS group
Procedure: ISO block — ISO block is a combined block of suprascapular nerve and brachial plexus cords using a single puncture
  Arms: ISO group

SUMMARY:
For shoulder analgesia, both ISO block and low volume scalene (LVS) block (using 5 ml of local anesthetics) are suggested to have a low incidence of hemi-diaphragmatic pariesis (HDP).

The aim of this study was to compare the incidence of HDP and the analgesic efficacy of the LVS block versus ISO block.

ELIGIBILITY:
Inclusion Criteria:

* patients who were scheduled for arthroscopic shoulder surgery

Exclusion Criteria:

* aged <18y
* BMI >35,
* ASA greater >III,
* an infection at the injection site
* has a contraindication for laryngeal mask or the medications used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
hemi-diaphragmatic pariesis | 2-4 hours
  diaphragmatic caudal displacement will be measured (in cm) with real time ultrasound before the block performance and after the procedure

SECONDARY OUTCOMES:
analgesic efficacy (block success) | 2-4 hours
  successful block = pain free (VAS 0) in recovery unit. VAS will be used to evaluate the pain (0 = pain free, 10= most sever pain)
patient satisfaction | 24 hours
  if the patient is satisfied with the analgesia technique or not
duration of analgesia | 24 hours
  duration between the block performance and the first requesting of pain killer (morphine)
total morphine dose | 24 hours
  the total morphine consumption within 24 hrs after the block performance

CONTACTS AND LOCATIONS:
Locations (1):
- Healthpoint Hospital, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taha AM, Yurdi NA, Elahl MI, Abd-Elmaksoud AM. Diaphragm-sparing effect of the infraclavicular subomohyoid block vs low volume interscalene block. A randomized blinded study. Acta Anaesthesiol Scand. 2019 May;63(5):653-658. doi: 10.1111/aas.13322. Epub 2019 Jan 30. PMID 30697688